## Informed consent

Belonging to: Validation of CPM#1 Compressibility in Healthy Volunteers in Rest and After Exercise

- I have read the information letter. I could ask questions which have been successfully answered.
- I have had enough time to decide whether I would participate at the investigation.
- I know participating is voluntary. I also know that I am able to decide on every moment to withdraw from the study. I am no obliged to say why I withdraw from the study.
- I give permission for the investigators to collect and use my data. The investigators will only use this to address and answer the study questions.
- I know that for inspection of the study some people will look into my data. Those
  persons are mentioned in the information letter. I give permission to these people to
  look into my data for inspection of the study.
- I want to participate at the study.

| My name is (participant): | |
|---|---|
| Autograph: | Date :// |
| I declare that I have informed the participant on the full extent of | |
| If there would become information known during the study which might influence the participant's informed consent, I will inform the participant on time. | |
| Name investigator (or representative): | |
| Autograph: | Date :// |

The participant will receive the full participant information flyer, together with a signed version of the informed consent form.